CLINICAL TRIAL: NCT01122108
Title: A Randomized, Single-Blind, Single Research Site, Comparison of Colesevelam Hydrogen Chloride (HCl) Powder For Oral Suspension Versus Generic Cholestyramine Through Use of the Bile Acid Sequestrant Acceptability (BASA) Scale in Generally Healthy Subjects
Brief Title: Comparison of Colesevelam Hydrogen Chloride (HCl) Powder For Oral Suspension Versus Generic Cholestyramine Through Use of the Bile Acid Sequestrant Acceptability (BASA) Scale
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Louisville Metabolic and Atherosclerosis Research Center (Other)
Collaborators: Provident Clinical Research (Other); Daiichi Sankyo (Industry)
Responsible Party: Harold Bays, MD, L-MARC Research Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2010-05-07; First posted 2010-05-13 (Estimated); Results first posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Bile Acid Sequestrant; Resin; Lipids; Glucose; Cholesterol; Diabetes Mellitus; Bile Acid Sequestrant Acceptability Scale
MeSH Terms: conditions — Diabetes Mellitus | interventions — Cholestyramine Resin; Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholestyramine 12 grams (Active Comparator): Cholestyramine 12 grams
  Interventions: Drug: Cholestyramine
- Colesevelam HCl (Active Comparator): Colesevelam HCl, 4 grams
  Interventions: Drug: Colesevelam HCl

INTERVENTIONS:
Drug: Cholestyramine — Cholestyramine 12 grams, one time dose
  Other Names: Questran
  Arms: Cholestyramine 12 grams
Drug: Colesevelam HCl — Colesevelam HCl, 4 grams, one time dose
  Other Names: Welchol
  Arms: Colesevelam HCl

SUMMARY:
The objective of this study is to compare the acceptability of Colesevelam HCl powder for oral suspension versus generic cholestyramine via the BASA scale, based upon an anticipated equivalent cholesterol lowering doses of each comparator drug.

DETAILED DESCRIPTION:
In 2009, colesevelam HCl was approved as a powder formulation. Little objective evidence exists comparing the acceptability of colesevelam HCl powder for oral suspension formulation versus other bile acid sequestrant powder formulations. A Bile Acid Sequestrant Acceptability (BASA) Scale was developed and validated as an instrument to compare the acceptability of different bile acid sequestrant preparations

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18-70 years of age
* In general good health (defined as study participants who are medically stable, meet protocol criteria, but who may also have non-exclusionary ongoing medical conditions).
* Subjects are capable of giving informed consent, or if appropriate, have an acceptable surrogate capable of giving consent on the subject's behalf.
* Subjects are willing and readily able to be contacted for post-study safety phone call assessments one to seven days after the single study visit.

Exclusion Criteria:

* Prior intolerance to bile acid sequestrants
* Known Phenylketonuria. Colesevelam (Welchol) for Oral Suspension contains 48 mg phenylalanine per 3.75 gram dose.
* Women who are either pregnant, or who are not practicing any form of birth control.
* Prior gastrointestinal surgery
* History of ongoing gastrointestinal symptoms (indigestion, constipation, or diarrhea)
* History of bowel obstruction, malabsorption, or irritable bowel syndrome
* History of esophageal disease
* Current or past history of gallbladder disease
* History of pancreatitis
* Subjects enrolled in another experimental (interventional) protocol within the past 30 days prior to visit 1.
* Diagnosis of diabetes mellitus
* Known history of triglyceride levels > 300 mg/dl.
* History of alcohol or drug abuse within 1 year of study entry
* Alcohol intake that exceeds more than 2 units of alcohol drinks per day
* Exposure to bile acid sequestrants (colesevelam HCl, cholestyramine, colestipol within 30 days of visit 1).
* Any other situation in which the Investigator makes the judgment that participation in the study would not be in the best interest of the study participant, or in the best interest of providing reliable study data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold E Bays, MD, Principal Investigator — L-MARC Research Center
Locations (1):
- L-MARC Research Center, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in April 2010 and ended in May 2010. Enrollment officially closed on May 24th, 2010. All patient screening and study visits were conducted at L-MARC Research Center's clinic.
Pre-assignment Details: Enrolled subjects were required to meet all of the inclusion and none of the exlusion criteria prior to being randomized to a group assignment. Subjects were also required to undergo vital sign obtainment, a brief physical exam, and a medical history review to ensure they were generally healthy.
Groups:
- Colesevelam HCl 3.75g First, Then Cholestyramine 12g: Colesevelam HCl 3.75g once orally in the first intervention and Cholestyramine 12g once orally in the second intervention. Both interventions were given on the same day, 30 minutes apart.
- Cholestyramine 12g First, Then Colesevelam HCl 3.75: Cholestyramine 12g once orally in the first intervention and Colesevelam 3.75g once orally in the second intervention. Both interventions were given on the same day, 30 minutes apart.
Period: Overall Study
Arm/Group | Colesevelam HCl 3.75g First, Then Cholestyramine 12g | Cholestyramine 12g First, Then Colesevelam HCl 3.75
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Colesevelam HCl (3.75g) vs Cholestyramine (12g): Although 2 different arms are used in this study, there is only one study group. All subjects received both treatment arms on the same day, just in varying orders. Thus, the participant flow and baseline characteristics are the same for both arms.
Arm/Group | Colesevelam HCl (3.75g) vs Cholestyramine (12g)
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 49.98 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Patient Acceptability of Colesevelam HCl Powder for Oral Suspension vs. Generic Cholestyramine Via the Bile Acid Sequestrant Acceptability (BASA) Scale, Based Upon an Anticipated Equivalent Cholesterol Lowering Doses of Each Comparator Drug.
Description: The bile acid sequestrant acceptability (BASA) scale has 4 scoring categories: taste, texture, appearance, and mixability. Participants rank each category separately. The best possible score for each category is 5, and the worst possible score for each category is 1.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: Units on BASA Scale
Groups:
- Colesevelam HCl (3.75g); Cholestyramine (12g): Although 2 different arms are used in this study, there is only one study group. All subjects received both treatment arms on the same day, just in varying orders. Thus, the participant flow and baseline characteristics are the same for both arms.
Arm/Group | Colesevelam HCl (3.75g) | Cholestyramine (12g)
Number analyzed (Participants) | 42 | 42
Units on BASA Scale
  Taste Score | 3.26 (.17) | 2.67 (0.18)
  Texture Score | 2.62 (0.19) | 2.36 (0.19)
  Appearance Score | 2.69 (0.12) | 3.48 (0.15)
  Mixability Score | 2.74 (0.14) | 2.6 (0.14)
Statistical Analysis 1: Comparison: Colesevelam HCl (3.75g) vs Cholestyramine (12g); The BASA scale was previously developed to effectively compare differing Bile acid sequestrant forumulations. The BASA scale should differentiate subject acceptability of Colesevelam HCl 3.75 vs Cholestyramine 12g based upon the sum of ratings for taste, texture, appearance and mixability. If normality hypothesis was rejected, then further inspection of the distribution utilizing normal quantile-quantile and kernel density plots was employed; Test type: Superiority or Other; p < 0.05, repeated measures analysis of variance — If a sequence was not found to be statistically significant, then that term was removed from final model. Normality of residuals was investigated for each outcome variable using the Shapiro-Wilk test; Sensitivity analyses were run to evaluate possible product by sequence interactions

2. Other Pre Specified Outcome: Weighted vs. Unweighted Composite BASA Scale Scores
Description: Aggregate scores were calculated for both the unweighted and weighted BASA scale scores for both Colesevlam HCL (3.75G) and Cholestyramine (12g). The best possible total BASA score is 20 and the worst possible total BASA score is 4. For the weighted version of the scale, the best possible total score is 60 and the worst possible total score is 4.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: Units on a BASA Scale
Arm/Group | Colesevelam HCl (3.75g) | Cholestyramine (12g)
Number analyzed (Participants) | 42 | 42
Units on a BASA Scale
  Total BASA Score | 11.31 (0.40) | 11.10 (0.43)
  Total Weighted BASA Score | 27.29 (1.21) | 26.05 (1.34)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed the informed consent to up to 7 days after the study visit.
Description: Adverse events were assessed in clinic during the study visit and through a follow-up phone call 1-7 days after the study visit.
Groups:
- More Than 30 Minutes After Last Beverage: This group summarizes the adverse events that occurred more than 30 mintures after the last beverage administered, and thus cannot be attributed to one specific bile acid sequestrant.
Arm/Group | Cholestyramine (12g) | Colesevelam HCl (3.75 Grams) | More Than 30 Minutes After Last Beverage
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 2/42 | 3/42 | 14/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cholestyramine (12g) (N=42) | Colesevelam HCl (3.75 Grams) (N=42) | More Than 30 Minutes After Last Beverage (N=42)
Belching (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Burping (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Throat (General disorders) | 1 (1) | 0 (0) | 0/32 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 1 (1)
Mild Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Mild Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gas (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Increased Urination (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Intermittent R Back Thigh Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Moderate Indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Severe Indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Moderate Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Used generally healthy subjects, for who lipid-altering medication may not be indicated; Compared the BAS on the same day; Evaluated estimated equal cholesterol lowering doses of each BAS, rather than same g amt of active drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes